CLINICAL TRIAL: NCT04843085
Title: Proteomic Characterization of Aggressive Oligodendrogliomas
Acronym: PROGLIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0074
Record Dates: First submitted 2020-12-17; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2020-12

CONDITIONS: Oligodendroglioma
Keywords: Oligodendroglioma; proteomic analysis; POLA network
MeSH Terms: conditions — Oligodendroglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumoral sample and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- O1: the more aggressive subgroup of oligodendroglioma samples of 30 patients
  Interventions: Other: Proteomic analysis
- O2: subgroup 2 of oligodendroglioma samples of 30 patients
  Interventions: Other: Proteomic analysis
- O3: subgroup 3 of oligodendroglioma samples of 30 patients
  Interventions: Other: Proteomic analysis
- IDH-mutant astrocytomas: patients with IDH-mutant astrocytomas, samples of 15 patients
  Interventions: Other: Proteomic analysis
- IDH-wildtype glioblastomas: patients with IDH-wildtype glioblastomas, samples of 15 patients
  Interventions: Other: Proteomic analysis

INTERVENTIONS:
Other: Proteomic analysis — : Proteomic analysis in the 3 subgroups of oligodendrogliomas (O1, O2 and O3) and in the comparator groups of IDH-mutant astrocytomas, IDH-wildtype glioblastomas and normal brain samples

SUMMARY:
Oligodendrogliomas represent a distinct subgroup of adult gliomas characterized by specific molecular alterations (1p/19q codeletion, mutations of IDH, TERT promoter, CIC, FUBP1). These tumors account for 5 to 10% of adult gliomas and are of special relevance in the neuro-oncology field because of their frequent chemosensitivity (Louis et al. 2016). The genetics of oligodendrogliomas is relatively well characterized but the mechanisms of oncogenesis for these tumors are poorly understood.

Although oligodendrogliomas prognosis is usually better than that of other adult glioma subtypes, it remains heterogeneous and there is no effective treatment at recurrence after radiotherapy and chemotherapy. Our recent work conducted within the INCa-funded national POLA network has related this clinical heterogeneity to inter-tumoral heterogeneity. Based on a transcriptomic analysis of a large series of oligodendroglial gliomas we identified 3 subgroups, the most aggressive group being characterized by aggressive clinical and molecular pattern. Recent studies, however, have shown a relatively low level of concordance between mRNA and protein expression, emphasizing the need to use proteomic-based approaches to better understand tumor biology. Taking advantage of the POLA cohort, we propose to expand our previous analysis by integrating a proteomic analysis of oligodendrogliomas.

The aim of this project is to identify drivers of oligodendroglioma subgroups, among which potential druggable targets (i.e receptors, metabolism effectors). For this purpose, the proteomic profiles of 90 oligodendrogliomas will be generated and integrated with transcriptomic, genomic and methylation profiles in order to identify signaling pathways specifically associated with each subtype, especially with the most aggressive one. Associations will be explored between candidate signaling pathways expression and clinical outcomes (survival, progression-free survival, objective response). The relevance of the 2 most promising candidate signaling pathways will be assessed in vitro and in vivo using genetically relevant mouse and xenograft models.

Our project will identify targetable oncogenic pathways associated with poor prognosis that could lead to new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* - transcriptomic (microarray) data available or possible to obtain them,
* methylation (450K) data available or possible to obtain them,
* genomic (SNP array) data available or possible to obtain them,
* sufficient material for proteomic analysis (frozen tumor samples)

Exclusion Criteria:

* opposed patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: samples of patients with oligodendrolioma, astrocytoma, glioblastoma and normal brain available in the POLA network biobank or the OncoNeuroTek tumor bank (Institut du Cerveau et de la Moelle Épinière)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
proteomic profiles | Baseline (at time of diagnosis surgery)
  Concordance of the classification of oligodendrogliomas based on their proteomic profiles with our previously identified oligodendrogliomas subgroups.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupement Hospitalier Est HCL, Bron
  - Institut du Cerveau et de la Moelle, Paris